CLINICAL TRIAL: NCT01573832
Title: Integrated Client Care Project Randomized Control Trial: Wound Care Evaluation
Brief Title: Integrated Client Care Project Trial: Wound Care Evaluation
Acronym: ICCP-WC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 11-289c
Record Dates: First submitted 2012-01-13; First posted 2012-04-10 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diabetic Foot Ulcer Intervention (Experimental)
  Interventions: Other: integrated client care group
- Diabetic Foot Ulcer Usual Care (No Intervention)
- Pionidal Sinus Ulcer Intervention (Experimental)
  Interventions: Other: integrated client care group
- Pionidal Sinus Ulcer Usual Care (No Intervention)

INTERVENTIONS:
Other: integrated client care group — receives integrated client care for wound treatment
  Arms: Diabetic Foot Ulcer Intervention; Pionidal Sinus Ulcer Intervention

SUMMARY:
This study will use a randomized control trial design to compare wound care clients who receive "integrated care" versus "usual care" in Community Care Access Centres (CCAC) in Ontario. Data will be collected by existing administrative databases and linked by the Institute for Clinical Evaluative Sciences (ICES). The researchers will analyze these databases and report findings.

DETAILED DESCRIPTION:
The researchers are interested in finding out whether the intervention ("integrated care") helps to improve patient outcomes. A randomized control trial of wound care clients in Ontario CCACs will show the effects of the intervention (integrated care) versus "usual care" clients. The researchers will also examine the financial system costs associated with providing "integrated care" to clients versus "usual care".

The researchers expect to answer the research question of whether there is difference in patient outcomes between "integrated care" versus "usual care clients." The researchers also would like to formulate a response for whether there will be financial system cost difference between "integrated care" and "usual care" clients.

The goal of this evaluation is to help decision-makers in the Ministry of Health and Long Term Care (MOHLTC), in the Community Care Access Centres (CCACs) and among provider organizations to improve the quality of care and patient outcomes for wound care clients, by evaluating innovations in the delivery of care.

ELIGIBILITY:
Inclusion Criteria:

* receives wound care from Community Care Access Centre provider
* adults over age 18 in Ontario

Exclusion Criteria:

* patients who do not receive wound care from Ontario Community Care Access Centres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13999 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients whose wound heals within the outcomes benchmark | 1 year
  percentage of patients whose wound heals within the outcomes benchmark

SECONDARY OUTCOMES:
time to wound healing outcomes | 1 year
  time to wound healing outcomes
total patient length of stay | at patient discharge, up to 365 days
  total patient length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Merrick F Zwarenstein, MB, PhD, Principal Investigator — Sunnybrook and Women's Hospital

REFERENCES:
- [Derived] Zwarenstein M, Shariff S, Mittmann N, Stern A, Dainty KN. A large cluster randomized trial of outcome-based pathways to improve home-based wound care. Trials. 2017 Aug 29;18(1):393. doi: 10.1186/s13063-017-2082-5. PMID 28851413